CLINICAL TRIAL: NCT02872831
Title: Prospective Randomized Study of Utilizing the 22-gauge Standard FNA Needle Compared to the SharkCore™ 22-gauge Fine Needle Biopsy (FNB) Needle in Patients With Solid Mass Lesions of the Gastrointestinal Tract
Brief Title: Beacon BNX™ Endoscopic Ultrasound (EUS)-Needle vs SharkCore™ Needle
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Departure from the institution
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15G.533
Record Dates: First submitted 2016-07-25; First posted 2016-08-19 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Cancer; Lymphadenopathy; Cholangiocarcinoma
Keywords: Fine needle aspiration
MeSH Terms: conditions — Pancreatic Neoplasms; Lymphadenopathy; Cholangiocarcinoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 22G SharkCore™ needle (Active Comparator): Covidien has recently released a novel SharkCore™ Fine Needle Biopsy (FNB) system for EUS-guided tissue acquisition of solid gastrointestinal lesions. With its unique bevel design, this needle has shown promising results to acquire histologic tissue as per oral communication with physicians around the country
  Interventions: Device: 22G SharkCore™ needle
- 22G BNX EUS-FNA needle (Active Comparator): The standard 22G BNX Endoscopic Ultrasound Fine needle aspiration (Beacon Endoscopic, Newton, MA) needle is routinely used for the evaluation of solid mass lesions in the pancreas and gastrointestinal tract.
  Interventions: Device: 22G BNX EUS-FNA Needle

INTERVENTIONS:
Device: 22G SharkCore™ needle — The 2 dedicated passes from the SharkCore™ needle will be placed in a jar with formaldehyde-based fixative and sent for routine histopathology evaluation. The cassette will be processed, embedded in paraffin, and then prepared in hematoxylin and eosin to be evaluated by one pathologist, who was blinded to the randomization sequence, for the presence of a histologic tissue. If adequate histologic tissue is present, the specimen will be graded as optimal or suboptimal.
  Arms: 22G SharkCore™ needle
Device: 22G BNX EUS-FNA Needle — Aspirates will be placed onto glass slides and preserved with Diff-Quik stain (American Scientific Products, McGraw Park, Illinois, USA). In addition, a smear will also be placed in alcohol for Papanicolaou staining. Any additional material was sprayed into Hanks's solution and sent for cell block processing. The cytology technician or cytopathologist on site will verify adequacy of specimens. At least two passes will be obtained from the lesion unless the technician established the presence of malignant appearing cells.
  Arms: 22G BNX EUS-FNA needle

SUMMARY:
The primary objective of this proposed prospective randomized, multi-center study is to evaluate the capability of the new 22G SharkCore™ needle to obtain tissue specimens and to compare its performance against the standard 22G BNX Endoscopic Ultrasound Fine needle aspiration (Beacon Endoscopic, Newton, MA) needle in the evaluation of solid mass lesions in the pancreas and gastrointestinal tract. The secondary objective is to determine the ability of the 22G SharkCore™ needle system to yield histologic tissue.

DETAILED DESCRIPTION:
Rationale:

A tissue core biopsy with preserved architecture is critical to diagnose and fully characterize certain neoplasms, such as lymphomas and GI stromal tumors (GIST). Moreover, tissue specimens for histologic examination also provides the opportunity to immunostain the tissue, further increasing differential diagnostic capabilities; reach a specific diagnosis for benign diseases not always obtainable with a cytological sample, thus sparing patients from more invasive and risky sampling procedures or costly and unnecessary follow-up examinations; perform tissue profiling and/or cell culture needed to guide targeted therapies for individualized treatment of patients with cancer of the GI tract.

There has previously been no needle available on the market that can accurately and consistently acquire EUS-guided histologic tissue from solid gastrointestinal lesions. Covidien has recently released a novel SharkCore™ Fine Needle Biopsy (FNB) system for EUS-guided tissue acquisition of solid gastrointestinal lesions. With its unique bevel design, this needle has shown promising results to acquire histologic tissue as per oral communication with physicians around the country (Douglas Adler and Christopher DiMaio).

Currently, there is no published clinical data on the capability of the SharkCore™ needle to obtain specimens via EUS guidance. The rationale of the currently proposed trial is to assess the operating characteristics SharkCore™ needle system and to determine the ability of this needle system to yield histologic tissue.

Medtronic Inc. has provided us with an unrestricted grant in order to evaluate the capability of the new 22G SharkCore™ needle to obtain tissue specimens and to compare its performance against the standard 22G BNX EUS-FNA.

Primary Objectives The primary objective of this proposed prospective randomized, multi-center study is to evaluate the capability of the new 22G SharkCore™ needle to obtain tissue specimens and to compare its performance against the standard 22G BNX Endoscopic Ultrasound Fine needle aspiration (Beacon Endoscopic, Newton, MA) needle in the evaluation of solid mass lesions in the pancreas and gastrointestinal tract. The secondary objective is to determine the ability of the 22G SharkCore™ needle system to yield histologic tissue.

Study Design We propose a prospective comparative study (22G SharkCore™ needle versus the 22G BNX EUS-FNA needle) randomized (randomization of the order of the needles) in crossover (on the same lesion) in samples of solid pancreatic and gastrointestinal tumors. Up to 6 sites in the United States will enroll the patients. The respective institutional investigators will review serious adverse events throughout the study. No interim analysis is planned.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will include anyone >18 years old that presents to the participating clinical institutions and requires an endosonographic evaluation for the presence of a solid-appearing mass lesion amenable to EUS access, and no contraindication to FNA as determined by standard clinical care

Exclusion Criteria:

1. Refusal to participate in the study
2. Solid-appearing mass lesion that in not amenable to EUS guided needle access for tissue acquisition
3. Patients with incomplete medical records
4. Pregnant patients
5. Prisoners
6. INR > 1.5
7. Platelets < 50,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the 22G SharkCore™ and the 22G BNX EUS-FNA needle | 12 months
  The primary endpoint measures of the study is to evaluate the diagnostic accuracy of the 22G SharkCore™ needle system or the 22G BNX EUS-FNA needle for the diagnosis malignancy in solid lesions of the pancreas and gastrointestinal tract. Diagnostic accuracy of the EUS needles for the diagnosis of malignancy is calculated as the number of True Positives with malignancy +True Negatives with malignancy/True Positives with malignancy +True Negatives with malignancy +False Positives with malignancy +False Negatives with malignancy.

SECONDARY OUTCOMES:
Sensitivity of the EUS Needles | 12 months
  Sensitivity is expressed in percentage and defines the proportion of true positive subjects with malignancy in a total group of subjects with malignancy.
Complications of the EUS Needles | 12 months
  Complications will be defined as any deviation from the clinical course after EUS-guided sampling as observed by the endosonographer or recovery suite nurse or as reported by patients. Excessive bleeding at the site of puncture, perforation, hypotension, and need for reversal medication will be documented.
Diagnostic sufficiency of Tissue obtained by the EUS Needles | 12 months
  Diagnostic sufficiency is defined as the proportion of patients in whom an on-site diagnosis was established within 2 passes of the EUS needles
Specificity of the 22G SharkCore™ needle and the 22G BNX EUS-FNA Needle for the diagnosis malignancy in solid lesions of the pancreas and gastrointestinal tract. | 12 months
  Specificity is defined as a proportion of subjects without the malignancy with negative test result in total of subjects without malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Ali Siddiqui, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No